CLINICAL TRIAL: NCT00460876
Title: Toxicity and Activity of Periocular Topotecan in Children With Retinoblastoma
Brief Title: Phase I Trial of Periocular Topotecan in Retinoblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital JP Garrahan (Other Government)
Responsible Party: Hospital JP Garrahan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14711603062
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Last update posted 2008-05-02 (Estimated); Status verified 2008-04

CONDITIONS: Retinoblastoma
Keywords: topotecan; periocular; chemotherapy
MeSH Terms: conditions — Retinoblastoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topotecan

SUMMARY:
This is a dose-escalation study aimed to assess the toxicity (and marginally the activity) of periocular topotecan in patients with relapsed-resistant retinoblastoma.

DETAILED DESCRIPTION:
Patients with bilateral retinoblastoma who have relapsed after attempts of conservative therapy with standard regimens such as carboplatin, etoposide, vincristine and external beam radiotherapy who face immediate enucleation of their single remaining eye are eligible for this protocol. Starting dose of topotecan will be 0.5 mg and dose escalation will be done by the accelerated titration method. Any Grade 3 ocular toxicity or grade 4 non ocular toxicity will be designed as the dose limiting toxicity. Grade 2 scleral toxicity will be considered for DLT. In case of grade 2 ocular toxicity or grade 3 systemic toxicity, the escalation dose will be 0.25 mg. Maximal dose will be 2 mg.

ELIGIBILITY:
Inclusion Criteria:

* Group Vb (Reese Ellsworth)
* Relapsed or progressed after carboplatin-based regimens and external beam radiotherapy
* Enucleation of the contralateral eye
* Normal renal and liver function

Exclusion Criteria:

* Presence of glaucoma, rubeosis iridis, anterior chamber extension
* Extraocular disease
* Adequate follow up impossible for social reasons

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity

SECONDARY OUTCOMES:
Response rate, description of toxicity, pharmacokinetic profile

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo L Chantada, MD, Principal Investigator — Hospital JP Garrahan
Locations (1):
- Hospital JP Garrahan, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Derived] Chantada GL, Fandino AC, Carcaboso AM, Lagomarsino E, de Davila MT, Guitter MR, Rose AB, Manzitti J, Bramuglia GF, Abramson DH. A phase I study of periocular topotecan in children with intraocular retinoblastoma. Invest Ophthalmol Vis Sci. 2009 Apr;50(4):1492-6. doi: 10.1167/iovs.08-2737. Epub 2008 Oct 31. PMID 18978345